CLINICAL TRIAL: NCT04418752
Title: Narrative Exposure Therapy for Traumatic Stress in Adults With Intellectual Disabilities: A Sequential Measurement Single Case Study Series
Brief Title: Narrative Exposure Therapy for Adults With Intellectual Disability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is no longer feasible due to the restrictions placed on access to potential participants during the COVID-19 pandemic.
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19101
Record Dates: First submitted 2020-05-07; First posted 2020-06-05 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: PTSD; Trauma, Psychological
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: The second phase of the research consists of a Sequential Measurement Single Case Study Series (SMSCSS) to explore the effectiveness of NET in reducing symptoms of traumatic stress in adults with ID. This requires measures to be completed at various time points across the research by both participants and carers. Inferences can then be made about changes in behaviour as a result of the therapy, particularly when a stable baseline has been established. In a naturalistic clinical setting, such as the current research, it is difficult to gain a stable baseline as the investigators would expect the potential for some change to occur in anticipation of the therapy. The investigators aim to collect three baseline measures prior to NET commencing; however, the investigators do not want to withhold therapy and risk attrition to obtain a stable baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological therapy (Other): Narrative Exposure Therapy will be delivered to all participants in the study except carer participants recruited to complete informant measures.
  Interventions: Other: Psychological therapy

INTERVENTIONS:
Other: Psychological therapy — The National Institute for Health and Care Excellence (2018) specifies NET as a psychological intervention for the treatment of PTSD or prominent symptoms of PTSD in adults. NET is a short-term treatment which incorporates elements of CBT exposure therapy and testimonial therapy. In exposure therapy, clients are encouraged to repeatedly discuss traumatic experiences in detail, including emotions and sensory experiences (Schauer, Elbert, & Neuner, 2011).Testimonial therapy involves "the construction of a detailed and coherent report of the survivor's biography including an explicit description of the traumatic events" (Neuner, Schauer, Roth & Elbert, 2002, pp.5-6). Therefore, NET aims to embed the traumatic experience within the context of the person's life and the mechanisms of change are theorised to be exposure and habituation to the traumatic experience and the reconstruction of autobiographical memory.

SUMMARY:
The purpose of the study is to identify how Narrative Exposure Therapy (NET) can be adapted for delivery with adults with mild Intellectual Disability (ID) and to explore whether NET can reduce symptoms of traumatic stress in this population.

The first phase of the research involves working with a speech and language therapist to make adaptations to the therapy and research materials for adults with mild ID. This work will then be triangulated by gaining feedback from a service user focus group on the accessibility of materials for adults with mild ID.

The second phase of the research consists of a 'sequential measurement single case studies series' to explore the effectiveness of Narrative Exposure Therapy (NET) in reducing symptoms of PTSD or prominent symptoms. Questionnaires will be completed before, during and after the therapy by both the adult with ID and a carer if possible and consenting. Electrodermal activity of participants will be measured throughout sessions (using an unobtrusive device) as an indicator of physiological arousal. All measures will be visually analysed using established criteria and statistical methods where possible. The impact of NET on a person's memory of events in their life will be explored by examining how coherent participants' accounts of traumatic experiences are before and after NET using coding systems developed by previous studies. An interview will take place approximately six weeks after therapy with the participant by an independent researcher. This will aim to collect qualitative data about the participants' experiences of NET and will be analysed using content analysis.

Participants will be recruited primarily from Intellectual Disability services in Nottinghamshire Healthcare NHS Foundation Trust. This will be extended to Derbyshire Healthcare NHS Foundation Trust and Lincolnshire Partnership NHS Foundation Trust if necessary (Secondary care). The investigators intend to recruit six participants and six carers to the study.

DETAILED DESCRIPTION:
People with ID have a substantially higher prevalence of mental health conditions when compared to the general population and are at greater risk of exposure to adverse life events. In a survey of 177 people with mild to moderate ID, 75% had experienced at least one traumatic event. It is therefore not surprising that, when compared to the general population, people with ID are more vulnerable to the development of post-traumatic stress disorder (PTSD).

Whilst the research suggests that people with ID have an increased risk of developing PTSD, there is a lack of research into trauma-focused interventions for this population. This is despite evidence that people with an ID within the mild range have been found to have the necessary skills to engage in the cognitive component of cognitive behavioural therapy (CBT) and the existence of a manual of CBT for people with mild ID and mood disorders.

The National Institute for Health and Care Excellence (NICE) recommends individual trauma-focused cognitive behavioural therapy (TFCBT) as a first line treatment for PTSD in adults and specifies Narrative Exposure Therapy (NET) as an example treatment. There appears to be no evidence to date of attempts to adapt NET for adults with ID and establish whether the therapeutic benefits described in the general population, in terms of reducing symptoms of trauma, are transferable to this population. This study would therefore be a first attempt in doing so.

The potential clinical benefit of the research is that a NICE recommended treatment for PTSD would be adapted for adults with mild ID and, if found to be effective, would increase the evidence base for trauma specific interventions for adults with ID. This would mean a better understanding of which therapies could help to reduce symptoms of traumatic stress in this population. At a service level, research into the effectiveness of different types of therapies guides best practice meaning resources are directed at therapies most likely to yield positive outcomes for service users.

The first phase of the research requires the lead investigator (Katie Marlow) to work with a speech and language therapist (SALT) to make general adaptations to the therapy and research materials for delivery with adults with mild ID. It is expected that the investigator and SALT will meet on multiple occasions. During these meetings, it is anticipated that:

* Feedback will be provided on the accessibility of the participant information sheets and consent forms for adults with mild ID.
* Adaptations will be made to the psychoeducation materials used within NET.
* Adaptations will be made to The Change Interview protocol.
* Advice will be offered on how NET sessions should be structured and delivered for adults with mild ID.

This work will be triangulated by a service user focus group (adults with ID) as patient public involvement (PPI) in the study design. Service users will be asked to provide feedback on the adaptations listed above in terms of accessibility for adults with mild ID. Changes will be made in line with this feedback and sent out again if necessary to gain further feedback. The investigators will ensure that adaptations do not lose fidelity with NET by using a fidelity framework informed by the NET manual. At this point it is likely that a substantial amendment will be submitted to the Research Ethics Committee to approve the adapted materials before use in the study.

The second phase of the research consists of a Sequential Measurement Single Case Study Series to explore the effectiveness of NET in reducing symptoms of traumatic stress in adults with ID. Participants will be recruited primarily from ID services in Nottinghamshire Healthcare NHS Foundation Trust. Recruitment will be extended to Derbyshire Healthcare NHS Foundation Trust and Lincolnshire Partnership NHS Foundation Trust if necessary. The initial approach will be from the Clinical Psychologist within the person's usual care team. Clinical Psychologists will be asked to explain and distribute the information sheet to potential participants on their caseload who meet the inclusion criteria. The information sheet will inform the potential participant of all aspects pertaining to taking part in the research. If the potential participant informs their Clinical Psychologist that they are interested in taking part, or would like to hear further information, the lead investigator will then contact the participant directly. If they subsequently agree to take part, they will be invited to attend an appointment with the investigator to complete a consent form. This will be at least one week after being given the information sheet. At this appointment, potential participants will be given opportunity to ask questions and invited to sign and date a written consent form prior to taking part in the study. The investigator will ask basic questions about the information sheet to check understanding and it will be recommended that a carer be present when they sign the consent form.

Participants must have capacity and capability to provide consent themselves due to the potentially distressing nature of trauma work, such as NET. Capacity to consent to the research will be assessed by the investigators following guidelines outlined in the Mental Capacity Act.

Once participants have consented to the research, the SALT and lead investigator will meet again to make specific adaptations to NET for the individual participant. This will involve accessing reports within participants' files, if given permission, such as the Wechsler Adult Intelligence Scale report and previous SALT reports. Following this, the lead investigator will deliver weekly sessions of NET, which have been adapted during the first phase of the research. This will be the equivalent of 12 sessions of NET and the investigators do not foresee each session lasting longer than one hour. NET is specified in NICE guidance for the treatment of PTSD in adults and therefore the participant is not receiving anything above usual treatment. Participants will be excluded from the research if they are already engaging in trauma-focused therapy with their Clinical Psychologist and no usual care will be withheld for the purposes of this study.

NET sessions will take place at clinic rooms within Nottinghamshire Healthcare NHS Foundation Trust; Horizon outpatients at Highbury Hospital and the Therapy and Treatment Centre in Mansfield (depending on the participant's preference). If participants are from within Derbyshire or Lincolnshire Trusts, more appropriate clinic space will be sought. All therapy sessions will be video recorded. This serves several purposes; to aid the investigator in the narration aspect of NET; to allow narratives of traumatic experiences to be compared before and after NET; to allow the investigators to complete observational measures of the participant; and to allow sessions to be quality assured by the Chief Investigator using a fidelity framework informed by the NET manual.

Participants will be asked to complete self-report measures prior to therapy (baseline), during therapy (at the start of each appointment) and after therapy (six weeks later). During therapy sessions, participants will be asked to wear an unobtrusive device (on two fingertips) to measure electrodermal activity as an indicator of their physiological arousal. The product works in conjunction with an apple/android device with the manufacturer's app installed; this device will be University of Nottingham owned.

Six weeks after completing NET, participants will be asked to take part in a change interview to gain their qualitative accounts of the therapy. The investigators will ask the Assistant Psychologist working within the ID service in Nottinghamshire Healthcare NHS Foundation Trust to conduct the interview given their experience working with adults with ID. If this is not possible, it will be conducted by an independent investigator from the Doctorate in Clinical Psychology programme; the interviewer will adhere to the same confidentiality procedures as the rest of the research team. The interview will take place at the same location where therapy was completed and will be audio recorded and subsequently transcribed by the lead investigator.

If the participant brings a carer to sessions, the participant will be encouraged to invite them into the initial psychoeducation session of NET to allow the carer to gain a greater understanding of the participant's trauma reactions and the potential utility of NET. The investigators will also encourage participants to invite their carer into the final part of therapy sessions for a debrief so that they are aware of the content covered and support which may be required following sessions.

Carers will also be asked for their participation in the research. If consenting, they will be asked to complete measures prior to therapy (baseline), at the end of therapy (final NET session) and at the change interview six weeks later. Within the participant consent form, participants are asked for their agreement for carers to complete questionnaires regarding their presentation. Carer participants will also have access to the information sheet for participants with ID so they are informed of all aspects of the research.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* 18 or over (no upper age limit due to ID services being lifelong).
* deemed to meet criteria for a mild intellectual disability, according to the clinical psychologist supporting recruitment.
* Experiencing traumatic stress, as assessed by their clinical psychologist using the Impact of Events Scale - Intellectual Disabilities. Traumatic stress will be a feature of their presenting problems but they are not required to have a diagnosis of PTSD (NET recommended to treat prominent symptoms also).
* English speaking.
* Able to travel to one of the therapy centres.
* Able to consent to the research, as assessed by both the clinical psychologist supporting recruitment and the student delivering NET.

Carer participants must be:

* 18 or over (no upper age limit).
* English speaking to undertake informant questionnaires.
* Able to comment on the symptoms of traumatic stress experienced daily by the participant.

Exclusion Criteria:

Participants will be excluded if they are:

* Substance dependent (NET requires participants to process traumatic experiences in detail; often substances are used as a way to block out these memories and therefore may impact on the therapy).
* Experiencing psychosis as assessed by both the clinical psychologist supporting recruitment and the student delivering NET.
* Currently an inpatient (NET at this time would be inappropriate due to challenging behaviour/level of illness).
* Currently engaging in a trauma-focused therapy with their psychologist (it would not be appropriate to interrupt potentially beneficial treatment).
* Currently engaging in other research projects (this would burden the participant and depending on the nature may affect results of this project).

Carer participants will be excluded if:

• They lack capacity to consent to take part in the research, as assessed by both the clinical psychologist supporting recruitment and the student delivering NET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change across the Impact of Events Scale-Intellectual Disabilities (IES-ID). | Through study completion, up to 24 weeks - at baseline, at each NET session and six weeks after NET has been completed.
  The IES-ID is a 22-item questionnaire scored on a three-point scale. It is designed for use with people with mild ID and measures symptoms of traumatic stress; higher scores indicate higher levels of traumatic stress. The authors found the scale to have excellent internal consistency, good to excellent test-retest reliability and good correlation with self-report measures of anxiety and depression.

SECONDARY OUTCOMES:
Change across the Clinical Outcome Routine Evaluation-Learning Disabilities (CORE-LD). | Through study completion, up to 24 weeks - at baseline, at each NET session and six weeks after NET has been completed.
  The CORE-LD is a 14-item questionnaire scored on a three-point scale for use with adults with ID receiving any form of psychological therapy; higher scores indicate higher levels of psychological distress. Within a sample of individuals with mild and moderate ID, the authors found the CORE-LD to be a valid measure with good test-retest reliability. The measure has been chosen as it captures general psychological distress and the unrevised version is widely used in NHS settings.
Change across the Lancaster and Northgate Trauma Scales - Informant Version (LANTS-IV). | Through study completion, up to 24 weeks - at baseline, at final session of NET and six weeks after NET has been completed.
  The LANTS-IV is a 43-item questionnaire completed by informants of adults with ID. It consists of a list of statements describing behaviours which may be exhibited by adults with ID who have experienced traumatic events. Informants are asked to rate each statement in terms of frequency on a six-point scale and severity on a three-point scale; higher scores indicate higher trauma related presentations. Within a sample of individuals with mild and moderate ID, the authors found the measure to have good internal reliability, test-retest reliability and construct validity. The LANTS-IV has been chosen as the investigators anticipate and encourage carer involvement in this research.

OTHER OUTCOMES:
Change across measures of Electrodermal activity (EDA) | Through study completion, up to 24 weeks - throughout baseline sessions, throughout each NET session and throughout session six weeks after NET has been completed.
  EDA will be measured using the Mindfield eSense Skin Response device - this measures skin conductance as an indicator of physiological arousal. Higher levels of EDA indicates higher levels of physiological arousal.
Change across the narrative cohesion of participants accounts of traumatic experiences | At the first and final session of NET - week 1 and week 12
  The narrative cohesion of participants accounts of traumatic experiences at the start and end of NET using coding systems developed by previous studies.

IPD SHARING:
Plan to Share IPD: No
Results will be written up in a peer-reviewed journal and as part of a Doctoral Thesis. Individual participant data will be anonymised. Should a request be made for individualised data, this would have to be approved by the various ethical and research boards involved.

REFERENCES:
- [Background] National Guideline Alliance (UK). Evidence reviews on care pathways for adults, children and young people with PTSD: Post-traumatic stress disorder: Evidence review J. London: National Institute for Health and Care Excellence (NICE); 2018 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK560231/ PMID 32757551
- [Background] Mevissen, L., Didden, R., & de Jongh, A. (2016). Assessment and treatment of PTSD in people with intellectual disabilities. Comprehensive guide to post-traumatic stress disorders, 281-299.
- [Background] Department of Health. (2005). Mental Capacity Act. Retrieved from https://www.legislation.gov.uk/ukpga/2005/9/pdfs/ukpga_20050009_en.pdf
- [Background] Hall JC, Jobson L, Langdon PE. Measuring symptoms of post-traumatic stress disorder in people with intellectual disabilities: the development and psychometric properties of the Impact of Event Scale-Intellectual Disabilities (IES-IDs). Br J Clin Psychol. 2014 Sep;53(3):315-32. doi: 10.1111/bjc.12048. Epub 2014 Mar 31. PMID 24684206
- [Background] Wigham S, Hatton C, Taylor JL. The Lancaster and Northgate Trauma Scales (LANTS): the development and psychometric properties of a measure of trauma for people with mild to moderate intellectual disabilities. Res Dev Disabil. 2011 Nov-Dec;32(6):2651-9. doi: 10.1016/j.ridd.2011.06.008. Epub 2011 Jul 12. PMID 21752595
- [Background] Brooks, M., Davies, S., & Twigg, E. (2013). A measure for feelings-using inclusive research to develop a tool for evaluating psychological therapy (Clinical Outcomes in Routine Evaluation-Learning Disability). British Journal of Learning Disabilities, 41(4), 320-329.
- [Background] Fletcher, R. J., Barnhill, J., McCarthy, J., & Strydom, A. (2016). From DSM to DM-ID. Journal of Mental Health Research in Intellectual Disabilities, 9(3), 189-204.